CLINICAL TRIAL: NCT05022680
Title: The Effects of Peer-led Walking Intervention With mHealth Technology for Physical Activity and Prenatal Health Outcomes
Brief Title: The Effects of Peer-led Walking Intervention With mHealth Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chin-Tsung Shen (Other)
Responsible Party: Sponsor-Investigator, Chin-Tsung Shen, head of administration, Mackay Medical College
Organization: Mackay Medical College (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LCF MOST 109-110
Record Dates: First submitted 2021-07-25; First posted 2021-08-26 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: mHealth Intervention
MeSH Terms: interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: randomize control trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants were used app to record their diet and steps every day (Experimental): Experimental group was the mHealth with peer led to improved their physical activity during pregnancy. Participants received app to record and monitor their physical activity every days and using it until childbirth.
  Interventions: Behavioral: mhealth
- non-mhealth (No Intervention): control group was the traditional prenatal care during pregnancy.

INTERVENTIONS:
Behavioral: mhealth — the peer-led intervention with mHealth technology (an application (APP) and Sports bracelet)
  Arms: Participants were used app to record their diet and steps every day

SUMMARY:
This study will apply the peer-led walking intervention with mHealth technology to maintain physical activity and promote prenatal health. Moreover, the participants of the trained peer mentors support women walking with mHealth technology, which has pregnant women using the APP to set goals, self-monitor, and self-manage, and it will continue to promote physical activity for overweight and obese pregnant women

DETAILED DESCRIPTION:
This study was to investigate the effectiveness of peer-led walking intervention with mHealth technology on physical activity, self-efficacy, weekly steps, exercise involvement and depression status. Participants of the trained peer mentors encourage women walking with mHealth technology, which has pregnant women using the APP to set goals, self-record, and self-monitor, and it will continue to promote physical activity for overweight and obese pregnant women.This study's results will be useful to healthcare providers who need to promote physical exercise and an active lifestyle for overweight and obese pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* women who had a pre-pregnancy body mass index of more than 25 kg/m2

Exclusion Criteria:

-

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 90 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
physical activity | throughout childbirth, average of 20-30 weeks
  physical activity (pregnancy physical activity questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Fang Lee, PhD, Principal Investigator — Mackay Medical College
Locations (1):
- Department of Nursing, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No